CLINICAL TRIAL: NCT06897800
Title: Correlations Between Cervial Pap Smear,Vaginal Microbiota, Human Papillomavirus and Index of Blood Vitamins and Metabolic Markers
Brief Title: Vaginal Microbiota and Its Association with Pap Smear Results, Human Papillomavirus, Vitamins, and Metabolic Mark
Status: Completed | Type: Observational
Sponsor: Cheng-Hsin General Hospital (Other)
Collaborators: Taipei Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: (803)109A-42
Record Dates: First submitted 2025-03-18; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Vaginal Microbiome
Keywords: vaginal microbiome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — vaginal discharge , cervical pap smear and blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The human microbiome, comprising bacteria, fungi, and viruses, plays a crucial role in host physiology, immune function, and disease susceptibility. While gut microbiota have been extensively studied, other sites, including the vaginal microbiome, exhibit distinct microbial compositions. The vaginal microbiome is typically dominated by Lactobacillus species, which contribute to vaginal health but fluctuate with hormonal changes, menopause, and metabolic factors.

This study analyzes the vaginal microbiome of 40 adult women using 16S rRNA sequencing and classifies them into Vaginal Community State Types (CSTs). CST IV, associated with dysbiosis, was most prevalent (55%). Postmenopausal women exhibited higher vaginal pH and increased CST IV prevalence (70%), while premenopausal women had more CST III (45%). SGLT2 inhibitor users showed higher beneficial CSTs (I, II) and lower CST IV.

Findings suggest strong links between vaginal microbiota, menopause, glycemic control, and antibiotic use, highlighting the need for targeted interventions to maintain vaginal health.

DETAILED DESCRIPTION:
Vaginal Microbiome, pH, Menopause, and Metabolic Factors

The human body is colonized by a vast array of symbiotic, commensal, and pathogenic microorganisms, including bacteria, fungi, and viruses. The relationship between these microorganisms and the host varies from mutualistic and commensal to pathogenic interactions, collectively referred to as the microbiome. The human microbiome resides on both external and internal surfaces of the body, playing a critical role in physiology, immune system development, digestion, and detoxification. The metagenome of bacterial populations within the human body contains at least 100 times more genes than the human genome, underscoring its crucial role in maintaining homeostasis and influencing disease pathogenesis.

The majority of bacterial communities reside in the gut, and over the past two decades, research has extensively focused on colonic microbiota, revealing intricate connections between gut microbes and various systemic physiological and pathological conditions. However, other anatomical sites, including the skin, oral cavity, urinary, and reproductive tracts, also host distinct microbial communities, which significantly differ from gut microbiota. The vaginal microbiome, in particular, is unique in that it is typically dominated by a single species of Lactobacillus, which is considered a hallmark of vaginal health. The composition of the vaginal microbiome is dynamic and changes across different life stages, influenced by hormonal fluctuations, menopause, metabolic factors, and external environmental factors.

This study employs 16S rRNA gene sequencing to comprehensively analyze the distribution of vaginal microbiota and their associations with lifestyle, metabolic conditions, and disease susceptibility, with the ultimate goal of optimizing women's health. Recent studies have increasingly adopted the classification of vaginal microbial communities using the concept of Vaginal Community State Types (CSTs), a framework proposed by Ravel in 2011. This study investigates the microbial composition of 40 adult female participants, categorizing their vaginal microbiomes into CST I, CST II, CST III, and CST IV.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the inclusion criteria

* Female participants
* History of sexual activity
* Age 30 years or older

Exclusion Criteria:

* Participants will be excluded from the study if they meet any of the following conditions:
* Currently pregnant at the time of enrollment or before sample collection day.
* History of total hysterectomy.

Ages: 32 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study participants will be selected from patients attending the Family Medicine outpatient clinic at Cheng Hsin General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Vaginal microbiome | Enrollment occurs at least 7 days before sampling. Participants must avoid menstruation, sex, douching, meds, and bathing within 24 hrs. All data collected in one visit within 2 hrs; study lasts within 2 weeks.
  The first swab of the vaginal secretion sample is tested for pH and glucose concentration using test strips in the clinic. The second swab is placed in a vial containing preservation solution. The label on the vial does not include the patient's name or medical record number but only indicates the sampling date and an identification number. The sample is temporarily stored at room temperature for one week in a lockable cabinet in the Family Medicine Department office. Subsequently, the sample is analyzed by a biotechnology company using mass cytometry and deep sequencing of bacterial 16S rRNA PCR to identify the various microbial communities present in the vaginal secretions.

SECONDARY OUTCOMES:
Cervical specimen | All data were collected during a single clinical visit within 2 hours, following vaginal discharge collection. The study period from enrollment to completion was approximately 2 weeks per participant.
  Participants underwent pelvic examination using an adjustable gynecological examination table. Disposable vaginal speculums and dedicated sampling swabs were used to ensure hygiene and standardization. Cervical cytology smears were interpreted by certified pathologists following the classification system provided by the Taiwan Health Promotion Administration. High-risk human papillomavirus (HR-HPV) genotyping included detection of HPV types 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, and 68.
blood, and urine samples | Blood and urine samples were collected on the scheduled sample collection day, prior to vaginal, and cervical specimen collection. All procedures were completed within 2 hours during the same clinical visit.Study duration was within 2 weeks.
  Participants underwent blood sampling after an 8-hour overnight fast for biochemical and nutritional assessments. The tests included complete blood count (CBC), white blood cell differential count, fasting blood glucose, glycated hemoglobin (HbA1c), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), triglycerides, C-reactive protein (CRP), vitamin A, vitamin D, vitamin E, vitamin B12, zinc, folate, serum iron, ferritin, total protein, albumin, and tumor marker CA125.
Anthropometric and Vital Measurements | Specimens were collected on the sample collection day, following completion of blood and urine sample collection. All procedures were completed within 2 hours during the same clinical visit.Study duration was within 2 weeks.
  Participants underwent anthropometric and Vital Measurements include height, weight, waist circumference, body fat percentage, and blood pressure values.
questionnaire | The questionnaire was completed post-exam on the sample day, in 10-15 minutes. All procedures finished within 2 hours. Study duration was within 2 weeks per participant.
  The questionnaire included items related to past medical conditions and vaccination history, current medication and supplement use, tobacco, alcohol, and betel nut use, dietary habits, menstrual cycle and sexual experience, and hygiene product usage patterns.

CONTACTS AND LOCATIONS:
Locations (1):
- Cheng Hsin General Hospital, Taipei, Taiwan, Taiwan